CLINICAL TRIAL: NCT01925742
Title: PEGASUS: PErsonalized Genomics for Prenatal Aneuploidy Screening USing Maternal Blood
Brief Title: Study of the Efficacy of New Non-invasive Prenatal Tests for Screening for Fetal Trisomies Using Maternal Blood
Acronym: PEGASUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Laval University (Other); Genome Canada (Other); Genome Quebec (Other); Genome British Columbia (Industry); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2014-1236; SIRUL-102531; B13-06-1236 (Other: Université Laval)
Record Dates: First submitted 2013-08-16; First posted 2013-08-20 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2016-04

CONDITIONS: Trisomy 21; Trisomy 18; Trisomy 13
Keywords: Fetal aneuploidy
MeSH Terms: conditions — Down Syndrome; Trisomy 18 Syndrome; Trisomy 13 Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Risk of aneuploidy (Experimental): Integrated prenatal screening for Down's syndrome (with follow-up fetal karyotype if positive); Serum QUAD Assay for aneuploidy screening; Semiconductor MPSS NIPT assay using ccfDNA in maternal blood; Optical-based MPSS NIPT assay using ccfDNA in maternal blood; Harmony™ Test (Ariosa Diagnostics)
  Interventions: Other: Integrated prenatal screening for Down's syndrome; Other: Serum QUAD Assay for aneuploidy screening; Other: Semiconductor MPSS NIPT assay using ccfDNA in maternal blood; Other: Optical-based MPSS NIPT assay using ccfDNA in maternal blood; Other: Harmony™ Test (Ariosa Diagnostics)
- High risk of aneuploidy (Experimental): Integrated prenatal screening for Down's syndrome (with follow-up fetal karyotype if positive); Serum QUAD Assay for aneuploidy screening; Semiconductor MPSS NIPT assay using ccfDNA in maternal blood; Optical-based MPSS NIPT assay using ccfDNA in maternal blood; Harmony™ Test (Ariosa Diagnostics) (subset)
  Interventions: Other: Integrated prenatal screening for Down's syndrome; Other: Serum QUAD Assay for aneuploidy screening; Other: Semiconductor MPSS NIPT assay using ccfDNA in maternal blood; Other: Optical-based MPSS NIPT assay using ccfDNA in maternal blood; Other: Harmony™ Test (Ariosa Diagnostics)

INTERVENTIONS:
Other: Integrated prenatal screening for Down's syndrome — Analysis of several serum biochemical markers, and fetal nuchal translucency by ultrasound, with computation of an individual risk of fetal aneuploidy.
  Other Names: IPS; Prenatal serum screening; Aneuploidy screening; Down's syndrome screening; Downs' syndrome screening
Other: Serum QUAD Assay for aneuploidy screening — Series of biochemical markers with results integrated into a computational estimate of risk of fetal aneuploidy
  Other Names: First trimester QUAD prenatal screening assay
Other: Semiconductor MPSS NIPT assay using ccfDNA in maternal blood — Analysis by next-generation sequencing of ccfDNA (circulating cell-free DNA) from maternal blood, using a targeted NIPT assay.
  Other Names: NIPD; MPSS; Non-invasive prenatal testing; Non-invasive prenatal diagnosis
Other: Optical-based MPSS NIPT assay using ccfDNA in maternal blood — Analysis by next-generation sequencing of ccfDNA (circulating cell-free DNA) from maternal blood, using an un-targeted NIPT assay.
  Other Names: NIPD; MPSS; Un-Targeted NIPD; Non-invasive prenatal testing; Non-invasive prenatal diagnosis
Other: Harmony™ Test (Ariosa Diagnostics) — Test that is commercially available (Ariosa Diagnostics). (will be used for benchmarking purposes in a subset of each arm)
  Other Names: DANSR Assay

SUMMARY:
Each year, 450,000 Canadian women become pregnant and, as a result of their participation in prenatal screening for Down syndrome, approximately 10,000 of them will have an amniocentesis (i.e. sampling of liquid surrounding the fetus) and of those, 315 will be found to carry a baby with Down syndrome and 70 normal pregnancies will be lost from complications of the procedure. It has been discovered recently that, during pregnancy, there is fetal DNA in maternal blood in sufficient quantities to be analysed and methods have been proposed to detect the presence or not of a fetus with Down syndrome using maternal blood. The introduction of genomic blood testing as proposed in the context of this project could lead to increased detection of Down syndrome, less invasive screening with 9700 amniocentesis avoided each year in Canada, improving the peace of mind of pregnant women, and preventing the accidental loss of 70 normal fetuses, at a lower overall cost than current practice. However, these methods still need to be validated before being appropriately introduced in routine care.

The study hypothesis is that new genomics-based non-invasive methods using fetal-DNA in maternal blood during pregnancy can be more effective than current prenatal screening methods for fetal aneuploidy.

This project will carry out an independent study that will validate the performance and utility of different new genomic technologies for screening in pregnant women using maternal blood. The team of researchers will compare the real-life performance of different non-invasive assays and strategies to screen for fetal aneuploidy, and identify an evidence-based cost-effective approach for implementation of this new technology in the Canadian health care system. The deliverables of this project will enable decision makers, pregnant women and their partner to make informed choices pertaining to prenatal genetic screening and diagnosis, such as screening for Down syndrome, and reduce the risk to pregnancies associated with amniocentesis.

DETAILED DESCRIPTION:
The present study is a real life comparative effectiveness study that will compare the performances and costs of several prenatal screening modalities for fetal aneuploidy (see interventions).

ELIGIBILITY:
Inclusion Criteria (High risk arm):

* women 19 years or older between 10 weeks and 23 weeks 6 days gestation undergoing amniocentesis or CVS for:
* positive prenatal screen;
* abnormal ultrasound
* previous pregnancy with trisomy
* patient or partner carrier of Robertsonian translocation involving chr 21
* positive NIPT result
* Maternal age 40 or more

Inclusion Criteria (Low risk arm):

* women 19 years and older who are 10 and 13 weeks 6 days gestation based on dating ultrasound (CRL) and are undergoing screening for Down syndrome (first trimester combined, SIPS or IPS)

Exclusion Criteria:

* women with multiple gestations
* women with twin demise (spontaneous or elective) at any gestational age
* women with active or history of malignancy

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3819 (Actual)
Dates: Start 2013-11; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Number of cases with Fetal trisomy 21, 18 or 13 | 6 weeks after the delivery date
  Only pregnant women will be recruited, fetal outcome will be assessed by fetal karyotype or at or after delivery.

SECONDARY OUTCOMES:
Number of women with assay failure | At end of pregnancy.

OTHER OUTCOMES:
Overall costs of screening algorithm | 6 weeks after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Francois Rousseau, MD MSc FRCPC, Principal Investigator — Universite Laval and CHU de Quebec; Sylvie Langlois, MD FRCPC, Principal Investigator — University of British Columbia
Locations (5):
- Canada (5):
  - Foothills Medical Centre, Calgary, Alberta
  - Children's & Women's Health Centre, Vancouver, British Columbia
  - The Ottawa Hospital, Ottawa, Ontario
  - CHU Ste-Justine, Montreal, Quebec
  - CHU de Québec, Québec, Quebec

REFERENCES:
- [Derived] Fibke C, Giroux S, Caron A, Starks E, Parker JDK, Swanson L, Jouan L, Langlois S, Rouleau G, Rousseau F, Karsan A. Effect of preexamination conditions in a centralized-testing model of non-invasive prenatal screening. Clin Chem Lab Med. 2021 Nov 11;60(2):183-190. doi: 10.1515/cclm-2021-0652. Print 2022 Jan 27. PMID 34761647
- [Derived] Rousseau F, Langlois S, Johnson JA, Gekas J, Bujold E, Audibert F, Walker M, Giroux S, Caron A, Clement V, Blais J, MacLeod T, Moore R, Gauthier J, Jouan L, Laporte A, Diallo O, Parker J, Swanson L, Zhao Y, Labelle Y, Giguere Y, Forest JC, Little J, Karsan A, Rouleau G. Prospective head-to-head comparison of accuracy of two sequencing platforms for screening for fetal aneuploidy by cell-free DNA: the PEGASUS study. Eur J Hum Genet. 2019 Nov;27(11):1701-1715. doi: 10.1038/s41431-019-0443-0. Epub 2019 Jun 23. PMID 31231136